CLINICAL TRIAL: NCT03481023
Title: Esophageal Cooling in Radiofrequency Cardiac Ablation: Pilot Study
Brief Title: Esophageal Cooling in Radiofrequency Cardiac Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riverside Medical Center (Other)
Collaborators: Attune Medical (Other)
Responsible Party: Principal Investigator, Brad Suprenant, Principal Investigator, Riverside Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMC # 186
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Esophageal Cooling Device; Radiofrequency Ablation; Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to which condition they were assigned; the Outcomes Assessor will be blinded to the hypotheses of the study as well as the condition to which the participant was assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Esophageal thermal regulation device (Experimental)
  Interventions: Device: EnsoETM
- LET monitoring (Active Comparator)
  Interventions: Procedure: Conventional Care

INTERVENTIONS:
Device: EnsoETM — Use of esophageal thermal regulation device during radiofrequency ablation.
  Arms: Esophageal thermal regulation device
Procedure: Conventional Care — Use of luminal esophageal temperature monitoring during radiofrequency ablation procedure.
  Other Names: LET monitoring
  Arms: LET monitoring

SUMMARY:
This pilot study evaluates the addition of the EnsoETM esophageal cooling device to the radiofrequency (RF) ablation procedure in the treatment of atrial fibrillation in adults. Half of participants will receive the EnsoETM in addition to RF ablation, while the other half will receive luminal esophageal temperature (LET) monitoring during RF ablation.

DETAILED DESCRIPTION:
Study Specific Procedures:

* Study specific imaging will include endoscopic evaluation of the esophagus one day before surgery at the time of the pre-op Transesophageal Echocardiography (TEE) and again 1-day post-op. This will include endoscopic esophageal intubation with visual assessment of the entire esophagus and grading of lesions. Coupled with this procedure will include endoscopic ultrasound assessment of the esophagus at the level of the left atrium with specific attention to the sub-mucosal layer that separates esophagus from the cardiac tissue. The patient will undergo moderate sedation during this procedure, which will accompany the TEE.
* The Esophageal Cooling Device (ECD) will be placed by trained study staff following endotracheal intubation. Proper positioning will be verified. A temperature probe will be placed to verify the patients core temperature. The target temperature will be set to the core temperature at the beginning of the procedure. Two minutes prior to ablation on the posterior wall the target temperature will be changed to the minimum temperature setting which will allow for maximal cooling. Cooling will take place throughout the duration of posterior wall ablation. After ablation in this territory is complete the target temperature will return to the patients core temperature. The device will be removed at the completion of the procedure by anesthesiology when there is no further need for an orogastric tube.
* LET monitoring will not be performed in the patients of the intervention group as the ECD is prohibitive. Therefore, ice lavage of the esophagus, as detailed below, will not be performed in this group.

Standard Care Procedures:

* Medical History will be obtained by interview and will involve identification of contraindications to the use of the ECD. This includes a history of esophageal perforation or varices. An allergy to silicone will be assessed.
* The patient's active medication list will be reviewed as is standard protocol for atrial fibrillation ablation, but this is not specific to the study as there are no medications that would impact the use of the ECD.
* All subjects will be on Protonix (40mg; twice daily) immediately following surgery for 30 days and anticoagulation for 3 months following surgery.
* The physical exam will be performed. Study specific exam is included as part of the airway assessment which is performed on a regular basis by anesthesiology. The oropharynx will be assessed prior to placement of the ECD.
* Radiofrequency ablation involving the posterior aspect of the left atrium will be performed with standard LET monitoring which may include intermittent boluses of iced lavaged saline through the nasogastric tube when the temperature rises above 1 degree centigrade. Termination of atrial fibrillation with provocation testing will be completed and further atrial tachyarrhythmia ablation will be carried out as indicated.
* The patient will follow-up in the office based on standard procedure with 10 day and 3 month follow-up to be scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Subject has an atrial arrhythmia requiring radiofrequency ablation on the posterior aspect of the heart.
* Subject is willing and able to provide informed consent.
* Subject is capable of adhering to the expectations of the study protocol (e.g., attending follow-up visit).

Exclusion Criteria:

* Subject has known esophageal deformity, or evidence of esophageal trauma.
* Subject has prior radiation therapy involving the esophagus.
* Subject has a history of esophageal disease (e.g., esophageal varices, cirrhosis, history of esophagectomy, previous swallowing disorders, or achalasia).
* Subject has ingested acidic or caustic poisons.
* Subject is incarcerated.
* Subject is pregnant or plans to become pregnant.
* Subject has a silicone allergy.
* Subject has esophageal bleeding prior to surgical procedure.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Riverside Medical Center, Kankakee, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No washout or run-in occurred after participants were enrolled in the study. Of the 7 patients that were recruited, one subject was excluded from the research study, because his BMI was outside of the study inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Esophageal Thermal Regulation Device | LET Monitoring
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esophageal Thermal Regulation Device | LET Monitoring | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 64.7 [58 to 70] | 61.3 [55 to 71] | 63 [55 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Baseline measure was collected via electronic chart review after informed consent was obtained and documented.
  Participants
    United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Esophageal Mucosal Damage
Description: Esophageal mucosal damage as assessed by endoscopic evaluation using Zagar's Modified Endoscopic Classification Scheme. Higher scores on this scale indicate a worse outcome. The grading system is as follows: Grade 0: Normal Examination; Grade 1: Edema and Hypermia of the Mucosa; Grade 2a: Superficial ulceration, erosions, friability, blisters, exudates, hemorrhages, whitish membranes; Grade 2b: Grade 2a pluse deep discrete or circumferential ulcerations; Grade 3a: Small scattered areas of multiple ulceration and areas of necrosis with brown-black or greyish discoloration; Grade 3b: Extensive necrosis. For this grading scale we used the following scoring:
  0=0 1=1 2a=2 2b=3 3a=4 3b=5
Time Frame: The post-intervention outcome measure was performed within 1 day after Pulmonary Vein Isolation.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Esophageal Thermal Regulation Device | LET Monitoring
Number analyzed (Participants) | 3 | 3
score on a scale | 1 [0 to 2] | 1.33333 [0 to 2]

2. Secondary Outcome: Number and Percentage of Participants With Treatment-Emergent Adverse Events [Safety and Adverse Events]
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Esophageal Thermal Regulation Device | LET Monitoring
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

3. Secondary Outcome: Presence of Esophageal Submucosal Damage, Indicated by Number of Ulcers as Assessed by Endoscopic Ultrasound (EUS)
Description: Altered submucosal tissue architecture as assessed by endoscopic ultrasound (EUS)
Time Frame: 1 day
Measure: Mean (Full Range); unit: Ulcers
Arm/Group | Esophageal Thermal Regulation Device | LET Monitoring
Number analyzed (Participants) | 3 | 3
Ulcers | .33 [0 to 1] | 1 [0 to 2]

ADVERSE EVENTS:
Time Frame: Adverse event monitoring was performed over the course of three months after the subject's surgery.
Description: There are no differences in the definition of adverse event or serious adverse event from the clinicaltrials.gov definition.
Arm/Group | Esophageal Thermal Regulation Device | LET Monitoring
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT03481023/Prot_000.pdf